CLINICAL TRIAL: NCT06912802
Title: Non-interventional Study to Assess the Impact of Myopia in Childhood and the Long-Term Complications in Adulthood on Health-Related Quality of Life (HRQoL).
Brief Title: Observational Survey Study on the Impact of Myopia and Its Complications on Quality of Life.
Status: Recruiting | Type: Observational
Sponsor: Santen SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: PMA-HEOR-QoL-001
Record Dates: First submitted 2025-03-17; First posted 2025-04-06 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Childhood Myopia: Parents (or other proxy) of children or adolescents aged 5 years or older suffering from myopia (low, moderate, or high myopia) defined by their refractive error;
  Interventions: Other: Non-Intervention
- Adulthood Myopia + Long-Term Complication: Adults suffering from myopia and its complications such as: cataract, macular degeneration, open-angle glaucoma, retinal detachment, and legal blindness/severe visual impairment.
  Interventions: Other: Non-Intervention

INTERVENTIONS:
Other: Non-Intervention — Non-Intervention study

SUMMARY:
This study aims to assess the impact of myopia in childhood and its long-term complications in adulthood on health-related Quality of Life (HRQoL), providing valuable data for cost-effectiveness models. It will gather country-specific information on healthcare resource utilization, including treatment costs, access to care, and reimbursement policies. In addition, the study will examine how myopia and its treatments affect daily activities and evaluate treatment satisfaction. No data on the efficacy of myopia treatments is collected in this study, and neither is the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Parents (or other proxy) of children or adolescents aged 5 years or older suffering from myopia (low, moderate, or high myopia) defined by their spherical equivalent (SER): Low myopia is from -0.5 D (inclusive) to -3.0 D (inclusive), Moderate myopia is from -3.0 D to -6.0 D (inclusive) and High myopia is <-6.0 D.
* Adults suffering from myopia and its complications such as: cataract, macular degeneration, open-angle glaucoma, retinal detachment, and legal blindness/severe visual impairment.
* Patients where myopia is a known or likely contributing factor to the complication.

Exclusion Criteria:

* Parents (or other proxy) of children aged 4 years and below.
* Patients where the complication is likely unrelated to myopia (e.g., cataract caused by diabetes) will be excluded

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children or adolescents aged 5 years or older suffering from myopia (low, moderate, or high myopia) and adults suffering from myopia and its complications such as: cataract, macular degeneration, open-angle glaucoma, retinal detachment, and legal blindness/severe visual impairment.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Group 1 respondents' assessment of EQ-5D-Y-3L (proxy) | Through study completion, an average of 6 months
  Group 1 respondents are parents (or other proxy) of children and adolescents suffering from myopia.
  The EQ-5D-Y-3L (European Quality of Life 5 Dimensions 3 Level) proxy version is an instrument used to assess health-related quality of life (HRQoL) of children and adolescents from the perspective of a parent, caregiver or another proxy. It uses a three-level scale (no problems, some problems or a lot of problems) along with a visual analogue scale (VAS) from 0 (worst imaginable health) to 100 (best imaginable health). The EQ-5D-Y-3L value sets will be used to calculate utility values.
Group 1 respondents' assessment of Bolt-on vision | Through study completion, an average of 6 months
  Group 1 respondents are parents (or other proxy) of children and adolescents suffering from myopia.
  The vision bolt-on assessment is an extension to the EQ-5D tool to specifically address the impact of vision impairment on a person's quality of life and consists of a single question in the same format.
Group 1 respondents' assessment of PedEyeQ (Pediatric Eye Questionnaire) | Through study completion, an average of 6 months
  Group 1 respondents are parents (or other proxy) of children and adolescents suffering from myopia.
  The PedEyeQ (Pediatric Eye Questionnaire) proxy version is a HRQoL (Health Related Quality of Life) assessment tool specifically designed to measure the impact of pediatric eye conditions on children. The tool consists of age-appropriate questionnaires (5-11 years old and 12-17 years old) that assess how vision problems affect daily activities, social interactions, school performance, and overall well-being of the child.
Group 2 respondents' assessment of EQ-5D-5L | Through study completion, an average of 6 months
  Group 2 respondents are adult patients suffering from myopia and a long-term complication of myopia.
  The EQ-5D-5L (European Quality of Life 5 Dimensions 3 Level) includes five questions covering mobility, self-care, usual activities, pain/discomfort and anxiety/depression. This questionnaire will be administered to adults suffering from myopia plus a complication. Each domain is rated from 1 (best quality) to 5 (worst quality), along with a VAS from 0 (worst imaginable health) to 100 (best imaginable health).
Group 2 respondents' assessment of Bolt-on vision | Through study completion, an average of 6 months
  Group 2 respondents are adult patients suffering from myopia and a long-term complication of myopia.
  The vision bolt-on is an extension to the EQ-5D tool to specifically address the impact of vision impairment on a person's quality of life. The EQ-5D-5L value sets will be used to calculate utility values for adults with myopia and its complications.
Group 2 respondents' assessment of NEI-VFQ-25 (National Eye Institute Visual Function Questionnaire-25) | Through study completion, an average of 6 months
  Group 2 respondents are adult patients suffering from myopia and a long-term complication of myopia.
  The NEI-VFQ-25 (National Eye Institute Visual Function Questionnaire-25) is a tool used to assess VRQoL (Vision Related Quality of Life) in individuals aged 18 and older. It consists of 25 items that measure the impact of vision impairment on daily activities and well-being across 12 domains, including visual function, mental health, social functioning, and role limitations. The NEI-VFQ-25 helps evaluate how visual problems affect a person's ability to perform tasks like reading, driving, and interacting socially.

CONTACTS AND LOCATIONS:
Locations (10):
- Copenhagen University Hospital, Copenhagen, Denmark
- University Hospital Necker Enfants Malades, Paris, France
- Germany (2):
  - Klinik für Augenheilkunde (Universitätsklinikum Freiburg), Freiburg im Breisgau
  - Universitäts-Augenklinik Mainz, Mainz
- Italy (2):
  - Meyer Children's Hospital IRCCS, Florence
  - Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Spain (2):
  - Estudio Oftalmologico, Madrid
  - The San Carlos Clinic Hospital (Hospital Clinico San Carlos-HCSC), Madrid
- St. Erik Eye Hospital, Solna, Sweden
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom